CLINICAL TRIAL: NCT06226051
Title: Growing Little PEAPODS Study: Association Between Prematurity and Body Composition, Nutrition Practices, and Neurodevelopmental Outcomes
Brief Title: Growing Little PEAPODS Study
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Meriter Hospital, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-0931; A536757 (Other: UW Madison); SMPH/PEDIATRICS/PEDIATRICS (Other: UW Madison); Protocol Version 9/11/2024 (Other: UW Madison); 2023-023 (Other: Meriter)
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Premature Birth; Premature Infant; Premature; Intrauterine Growth Restriction; Small for Gestational Age at Delivery
MeSH Terms: conditions — Premature Birth; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PEAPOD device: Premature babies will be evaluated using the PEAPOD Infant Body Composition measuring device
  Interventions: Device: PEAPOD Infant Body Composition measuring device

INTERVENTIONS:
Device: PEAPOD Infant Body Composition measuring device — PEAPOD is a device to that collects body composition measurements.

SUMMARY:
The goal of this clinical trial is to learn more about how the food and nutrition babies receive while in the Neonatal Intensive Care Unit (NICU) influences their ability to gain weight and fat-free mass, and their future growth and development.

Participants will:

* have body growth measurements collected using the PEAPOD device
* have nutritional information collected, and
* be followed for neurodevelopmental outcomes

Participants can expect to be in the study for 36 months.

ELIGIBILITY:
Neonate Inclusion Criteria:

* Born inpatient at Meriter Hospital, Inc. at or above 22 gestational weeks. Upper limit is 32 weeks 6 days GA (possible gestational age range from 22w0d-32w6d)

Neonate Exclusion Criteria:

* Known genetic condition that impacts neurodevelopmental outcomes or brain structure development
* Multiple major congenital anomalies
* Per the investigator's opinion, the subject will likely require transfer to American Family Children's Hospital (AFCH) before 36 weeks PMA

  * Any neonate who enrolls in the study and then unexpectedly requires transfer to AFCH before 36 weeks PMA will be excluded from the study if they are unable to obtain at least one body composition measurement before transfer. Body composition data points can only be collected at Meriter Hospital due to the location of PEAPOD

Birthing Parent Inclusion Criteria:

* Birthing parent must speak English or Spanish due to consent documents
* Able to understand and willing to sign a written informed consent document
* Primary caregiver of a neonate who is eligible to participate in the study
* Agrees to enroll neonate into the study
* Willing to comply with all study procedures and be available for the duration of the study
* Age 15 or older

Birthing Parent Exclusion Criteria:

* Subject is unable to provide informed consent, including subjects in foster care and subjects within state custody
* Does not plan to maintain custody of the child after birth, such as in instances of adoption or surrogacy

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 120 neonates born inpatient at Meriter Hospital, Inc. ≤ 32 weeks 6 days (32w6d) GA (possible gestational age range from 22w0d-32w6d)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the correlation between nutritional intake over the first two weeks of life and the percent increase in fat-free mass measured by the PEAPOD | Birth to 2 weeks
  The least absolute shrinkage and selection operator technique will be utilized to determine whether fat intake predicts a percent increase in fat-free mass
To evaluate the correlation between higher nutritional intake in the first 2 weeks of life and the General Movement Assessment (GMA) and/or the Bayley Scales of Infant and Toddler Developmental Scores (Bayley) | Birth to 36 months
  The least absolute shrinkage and selection operator technique will be utilized to determine whether higher nutritional intake predicts Bayley cognitive scores
To evaluate the correlation between the percent increase in fat-free mass and the GMA and/or Bayley scores. | Birth to 36 months
  The least absolute shrinkage and selection operator technique will be utilized to determine whether the percent increase in fat-free mass predicts GMA scores and Bayley scores.

CONTACTS AND LOCATIONS:
Overall Officials: Whitley Hulse, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Meriter Hospital, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No